CLINICAL TRIAL: NCT00856674
Title: A Dose-Escalating Phase I Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Intravenous OPL-CCL2-LPM in Patients With IgA Nephropathy
Brief Title: Safety Study of of Intravenous CCL2-LPM in Patients With IgA Nephropathy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to resources and slow enrollment; not due to safety
Sponsor: Osprey Pharmaceuticals USA, Inc. (Industry)
Responsible Party: Barbara K. Finck, M.D., Senior Vice President and Chief Medical Officer, Osprey Pharmaceuticals USA, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPL01-CCL2
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-06

CONDITIONS: IGA Nephropathy; Proteinuria
Keywords: IgA nephropathy; chemokine fusion protein; leukocyte population modulator; phase-1
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: OPL-CCL2-LPM — CCL2-LPM
  intravenous 0.001 mg/kg, 0.01 mg/kg, 0.05 mg/kg, 0.1 mg/kg, 0.5 mg/kg, 1 mg/kg
  2 doses one week apart
  Other Names: CCL2-LPM; CCL2-SA1 fusion protein

SUMMARY:
The purpose of this study is to evaluate the safety of several dose levels of CCL2-LPM in patients with IgA Nephropathy who have high levels of protein in the urine.

DETAILED DESCRIPTION:
In spite of adequate blood pressure control and diet, 30 percent of patients with IgA nephropathy continue to secrete large amounts of protein in the urine and have a high likelihood of progressing to end-stage renal disease over 5-10 years and eventually requiring dialysis or kidney transplant. In IgA nephropathy, the injured kidney tissue secretes a messenger that recruits white blood cells (leukocytes) into the kidney. This messenger is the chemokine, CCL2. As a consequence CCL2 also is excreted into the urine and can be measured as evidence of inflammation in the kidney. This study evaluates the safety of a new potential therapy,CCL2-LPM (leukocyte population modulator), for IgA nephropathy. CCL2-LPM is composed of the messenger chemokine, CCL2, fused to an enzyme that inhibits protein production by the leukocytes and prevents the leukocytes from migrating into the kidney. The CCL2 end of the molecule targets only a small subset of leukocytes that have the corresponding receptor for CCL2 on the surface. After CCL2 binds to its receptor it is drawn inside the cell and carries the enzyme into the cell. The targeted cells are prevented from entering the kidney and causing further damage. Thus, CCL2-LPM may interrupt the ongoing cycle of inflammation that leads to end-stage renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven IgA nephropathy
* GFR > 30 mL/min
* Urinary protein > 700 mg/day
* Stable serum creatinine
* Urine CCL2/creatinine > 250 pg/mg
* Stable doses of medications
* ACEI and/or ARB maximized to control hypertension and proteinuria

Exclusion Criteria:

* Other causes of nephropathy
* Pregnant or nursing females
* Prednisone > 10 mg/day
* Other prohibited medications
* BP > 140/90
* BMI > 35
* Concurrent infection requiring treatment
* Clinical significant concurrent medical conditions
* Known allergy or sensitivity to formulation ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | 30 days after last dose of study drug

SECONDARY OUTCOMES:
Pharmacokinetics: urine protein/creatinine, urine CCL2/creatinine, sCRP change, change in leukocyte subsets by flow cytometry analysis | over 30 day period

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Pichette, M.D., Ph.D., Principal Investigator — Hopital Maisonneuve-Rosemont, Univeristy of Montreal; Michelle Hladunewich, M.D., Principal Investigator — Sunnybrook Health Sciences Centre; Bryan Curtis, M.D., Principal Investigator — Eastern Health, HSC, Memorial University
Locations (3):
- Canada (3):
  - Eastern Health, HSC, Memorial University, St. John's, Newfoundland and Labrador
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hoptial Maisonneuve-Rosemont, Montreal, Quebec

REFERENCES:
- [Background] McDonald JR, McManaman JL, Yong VW. The therapeutic potential of chemokine-toxin fusion proteins. IDrugs. 2001 Apr;4(4):427-42. PMID 16015483
- [Background] Eardley KS, Zehnder D, Quinkler M, Lepenies J, Bates RL, Savage CO, Howie AJ, Adu D, Cockwell P. The relationship between albuminuria, MCP-1/CCL2, and interstitial macrophages in chronic kidney disease. Kidney Int. 2006 Apr;69(7):1189-97. doi: 10.1038/sj.ki.5000212. PMID 16609683
- [Background] McIntosh LM, Barnes JL, Barnes VL, McDonald JR. Selective CCR2-targeted macrophage depletion ameliorates experimental mesangioproliferative glomerulonephritis. Clin Exp Immunol. 2009 Feb;155(2):295-303. doi: 10.1111/j.1365-2249.2008.03819.x. Epub 2008 Nov 25. PMID 19040610
- [Background] Reich HN, Troyanov S, Scholey JW, Cattran DC; Toronto Glomerulonephritis Registry. Remission of proteinuria improves prognosis in IgA nephropathy. J Am Soc Nephrol. 2007 Dec;18(12):3177-83. doi: 10.1681/ASN.2007050526. Epub 2007 Oct 31. PMID 17978307
- [Background] Morii T, Fujita H, Narita T, Koshimura J, Shimotomai T, Fujishima H, Yoshioka N, Imai H, Kakei M, Ito S. Increased urinary excretion of monocyte chemoattractant protein-1 in proteinuric renal diseases. Ren Fail. 2003 May;25(3):439-44. doi: 10.1081/jdi-120021156. PMID 12803507
- [Background] Rovin BH. The chemokine network in systemic lupus erythematous nephritis. Front Biosci. 2008 Jan 1;13:904-22. doi: 10.2741/2731. PMID 17981599
- [Background] Nair R, Walker PD. Is IgA nephropathy the commonest primary glomerulopathy among young adults in the USA? Kidney Int. 2006 Apr;69(8):1455-8. doi: 10.1038/sj.ki.5000292. PMID 16531983